CLINICAL TRIAL: NCT00942955
Title: A Randomized Controlled Multi-center Trial of a Point-Of-Care Chemistry Test for Reduction of Turnaround and Clinical Decision Time in the Emergency Department
Brief Title: Point-Of-Care Chemistry Test (POCT) Effect on the Emergency Department (ED)
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Shin Sang Do/Assistant professor, Seoul National University Hospital Department of Emergency medicine
Other Study IDs: SNUEMS200801
Record Dates: First submitted 2009-07-20; First posted 2009-07-21 (Estimated); Last update posted 2009-07-21 (Estimated); Status verified 2009-07

CONDITIONS: Emergency Department; Length of Stay; Turnaround-time
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- CLT: The patients whose blood are analyzed by conventional central laboratory.
- POCT: the patients group whose lab analyze by POCT device.

SUMMARY:
The hypothesis of this study is that POCT will shorten ED turn-around-time (TAT) such as blood drawing TAT, lab TAT, and decision TAT.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 15 years
* clinically required to have chemistry lab tests
* agreement

Exclusion Criteria:

* no agreement
* ESI level 1

Min Age: 15 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: This study was performed in five EDs. Three were urban EDs with 30,000 to 45,000 annual visits, and two were suburban EDs with 15,000 to 25,000 annual visits. Each hospital has its own central laboratory which can test the same emergency chemistry tests, including liver panel (alkaline phosphatase, protein, albumin, total bilirubin, direct bilirubin, GOT, and GPT), renal panel (BUN, creatinine, calcium, and phosphorus), pancreas enzymes (amylase, lipase), electrolytes (sodium, potassium, chloride, total CO2), lipid panel (total cholesterol, triglyceride, LDL-cholesterol, HDL-cholesterol), and blood gases (pH, pO2, pCO2, and bicarbonate).
Sampling Method: Probability Sample
Dates: Start 2009-01; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)